CLINICAL TRIAL: NCT06899945
Title: The Effects of Vibration Therapy at Different Frequencies on Pain, Range of Motion, Functionality, Joint Position Sense, and Quality of Life in Individuals With Rotator Cuff Syndrome
Brief Title: Effects of Vibration Frequencies in Rotator Cuff Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Emre DANSUK, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-1958
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Rotator Cuff Syndrome; Vibration Therapy
Keywords: Rotator Cuff Syndrome; Vibration Therapy; Pain; Functionality; Proprioception; Quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Conventional Physiotherapy) (Active Comparator): Participants in the control group will receive only conventional physiotherapy without vibration therapy. This ensures a baseline comparison to assess the effectiveness of vibration therapy.
  Treatment Modalities:
  TENS therapy (20 minutes, 100 Hz) Mobility exercises (wand exercises, Codman exercises, active/passive stretching) Strengthening exercises (theraband-based training) Frequency: 5 sessions per week Total Treatment Period: 3 weeks
  Interventions: Other: conventional physiotherapy program
- Vibration Therapy (16.7 Hz) Group (Experimental): This group will receive vibration therapy at 16.7 Hz using a percussion massage gun (Hypervolt device (Hyperice, CA, USA)) along with a standard physiotherapy program. The treatment protocol mirrors the 33 Hz group, except for the vibration frequency.
  Duration: 3 minutes per muscle Frequency: 3 times per week Total Treatment Period: 3 weeks Additional Treatment: Standard physiotherapy (TENS, mobility exercises, and strengthening)
  Interventions: Device: a percussion massage gun (Hypervolt device (Hyperice, CA, USA)); Other: conventional physiotherapy program
- Vibration Therapy (33 Hz) Group (Experimental): Participants in this group will receive vibration therapy at 33 Hz using a percussion massage gun (Hypervolt device (Hyperice, CA, USA)) in addition to a standard physiotherapy program. The therapy will target the deltoid, supraspinatus, infraspinatus, and teres minor muscles, applying vibration along the origin-insertion pathway.
  Duration: 3 minutes per muscle Frequency: 3 times per week Total Treatment Period: 3 weeks Additional Treatment: Standard physiotherapy (TENS, mobility exercises, and strengthening)
  Interventions: Device: a percussion massage gun (Hypervolt device (Hyperice, CA, USA)); Other: conventional physiotherapy program

INTERVENTIONS:
Device: a percussion massage gun (Hypervolt device (Hyperice, CA, USA)) — Vibration application will be applied to the individuals in this group in addition to conventional methods. Vibration application will be applied to the deltoid, supraspinatus, infraspinatus, and teres minor muscles with a percussion massage gun (Hypervolt device (Hyperice, CA, USA)) along the origo-insertio line for 3 minutes for each muscle group. Vibration application will be performed using the soft head of the percussion massage gun. Vibration therapy will be applied 3 days a week for 3 weeks.
  Arms: Vibration Therapy (16.7 Hz) Group; Vibration Therapy (33 Hz) Group
Other: conventional physiotherapy program — Participants in the conventional physiotherapy program will follow a 3-week exercise plan, with sessions 5 days per week, each lasting 30 minutes under physiotherapist supervision.
  Treatment includes:
  TENS therapy (20 min, 100 Hz) on the painful area. Wand exercises for flexion, abduction, extension, internal, and external rotation (10 reps/set).
  Codman exercises for flexion, abduction, and circular movements (10 reps/set). Active & passive stretching for flexion, abduction, internal, and external rotation (10 reps/set).
  Finger ladder exercises for flexion and abduction (10 reps/set). Strengthening with a theraband for flexion, abduction, external/internal rotation, and extension, adjusted based on progress (10 reps/set).
  This exercise program will be applied to all study groups.

SUMMARY:
This study aims to investigate the effects of vibration therapy applied at different frequencies using a percussion massage gun on pain, range of motion (ROM), functionality, joint position sense, and quality of life in individuals with rotator cuff syndrome.

Rotator cuff syndrome is a common shoulder disorder caused by excessive use, muscle weakness, trauma, or instability, leading to pain, restricted movement, and reduced functional capacity. Although percussion massage therapy has gained popularity for its potential therapeutic benefits, there is limited scientific evidence on its effectiveness in improving ROM, pain reduction, and functional outcomes.

A total of 48 participants diagnosed with rotator cuff lesions will be included in the study and divided into three groups:

Vibration Group (33 Hz) Vibration Group (16.7 Hz) Control Group (Conventional Physiotherapy)

The intervention will include:

Conventional physiotherapy exercises applied to all groups, Vibration therapy with a percussion massage gun applied to the experimental groups, targeting the deltoid, supraspinatus, infraspinatus, and teres minor muscles for three minutes per muscle, three times per week for three weeks.

Outcome Measures:

Pain: Visual Analog Scale (VAS) ROM & Joint Position Sense: Measured using the Goniometer Pro mobile application Functionality: Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire Quality of Life: Rotator Cuff Quality of Life (RC-QoL) questionnaire

Hypotheses:

Vibration therapy at different frequencies will significantly impact pain, ROM, functionality, joint position sense, and quality of life.

33 Hz vibration therapy will be more effective than 16.7 Hz in improving outcomes.

The data will be analyzed using SPSS 25, with statistical tests applied based on data distribution. This research aims to contribute to the understanding of vibration therapy's role in managing rotator cuff syndrome and its effectiveness in clinical rehabilitation.

DETAILED DESCRIPTION:
Rotator cuff syndrome is a common shoulder disorder caused by excessive use, muscle weakness, trauma, or instability. It often results in pain, restricted movement, and reduced functional capacity. The condition is associated with subacromial space compression, leading to tendinitis, partial tears, or full rupture, which affects daily activities and overall quality of life.

Percussion massage therapy is an emerging treatment method that combines elements of traditional massage and vibration therapy. Introduced in the 1950s by Robert Fulford, it was later developed into handheld devices for self-administered and professional use. Percussion therapy is believed to reduce pain, enhance circulation, improve tissue healing, decrease muscle spasms, and increase joint range of motion (ROM).

However, scientific evidence regarding its effectiveness, particularly in rotator cuff syndrome, remains limited. This study aims to investigate the effects of different frequencies of vibration therapy applied with a percussion massage gun on pain, ROM, functionality, joint position sense, and quality of life in individuals with rotator cuff syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with rotator cuff lesion,
* Experiencing shoulder pain for at least 3 weeks,
* Aged between 30-60 years,
* Having restricted shoulder range of motion.

Exclusion Criteria:

* Individuals with an additional orthopedic or neurological disorder affecting the shoulder,
* Those with a history of previous shoulder trauma,
* Individuals who have participated in a physiotherapy program within the last 3 months,
* Those unable to tolerate vibration therapy.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of Joint Position Sense | 3 weeks
  The joint position sense of the participants in the study will be measured using the Fizyosoft Extremity ROM system. Joint position sense will be evaluated in 60-degree shoulder flexion and abduction movements.
  Participants will be asked to lift their arm to 60 degrees with their eyes open and remember the position. Then, they will be instructed to replicate the same movement with their eyes closed. The shoulder angle will be measured while their eyes are closed.
  The difference between the open-eye and closed-eye measurements will be recorded as the joint position sense. This method will be applied at 60-degree shoulder flexion and abduction .The average of two trials will consider for data evaluation.

SECONDARY OUTCOMES:
Visual Analogue Scale | 3 weeks
  Visual Analogue Scale (VAS) will be used to evaluate the pain intensity of patients. VAS consists of a 10 cm long horizontal line. '0' represents no pain, '10' represents unbearable pain. During our evaluation, patients will be asked to mark the level of pain they feel on this chart, and the distance to the starting point will be measured and recorded with the ruler.
Range of Motion | 3 weeks
  The shoulder range of motion (ROM) of the participants included in the study will be measured using the Fizyosoft Extremity ROM system.
  The measurements will be recorded as follows:
  Flexion and abduction: 0-180 degrees Internal and external rotation: 0-90 degrees.
Disabilities of the Arm, Shoulder, and Hand Questionnaire | 3 weeks
  The DASH questionnaire is used to assess physical disability and functionality in upper extremity injuries. It consists of three subcategories:
  The first section contains 30 questions measuring functional and symptom scores, including:
  21 questions evaluating daily living activities, 5 questions assessing symptoms (pain, activity-related pain, tingling, weakness, and movement restriction), 4 questions related to social function, work, sleep, and self-confidence. The work module consists of 4 additional questions, evaluating the participant's ability to perform work-related tasks.
  Each question is answered using a 5-point Likert scale:
  1. = No difficulty
  2. = Mild difficulty
  3. = Moderate difficulty
  4. = Severe difficulty
  5. = Unable to perform the activity A higher total score indicates a greater level of disability.
Assessment of Quality of Life | 3 weeks
  The Rotator Cuff Quality of Life (RC-QoL) questionnaire was developed by Hollishead et al. and was validated for the Turkish population by Çınar-Medeni et al. in 2015. This questionnaire is a specific assessment tool designed to evaluate the quality of life in individuals with rotator cuff pathology.
  The scale consists of 34 questions categorized into five sections:
  Physical symptoms Work-related activities Daily living activities Social aspects Emotional well-being
  Each question is scored on a scale from 0 to 100, where:
  0 = Severe pain or impairment 100 = No pain or impairment A higher score indicates better quality of life. The total score is calculated by summing the scores of the answered questions, dividing by the number of answered questions, and converting the result into a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Dansuk, PhD, Principal Investigator — Medipol University
Locations (1):
- Emre Dansuk, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No